CLINICAL TRIAL: NCT05575076
Title: An Open-label, Long-term Extension Study to Evaluate the Safety and Tolerability of Simufilam 100 mg Tablets in Participants With Mild to Moderate Alzheimer's Disease
Brief Title: Open-label Extension for Phase 3 Clinical Trials of Simufilam
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Cassava Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTI-125-10
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Simufilam

STUDY DESIGN:
Intervention Model Description: Open-label extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Simufilam 100 mg (Experimental): simufilam 100 mg oral tablet, twice daily
  Interventions: Drug: Simufilam

INTERVENTIONS:
Drug: Simufilam — simufilam 100 mg oral tablet, twice daily
  Other Names: PTI-125

SUMMARY:
The goal of this open-label extension study is to assess long-term safety and tolerability of simufilam 100 mg in subjects who have completed the RETHINK-ALZ or REFOCUS-ALZ Phase 3 clinical trials.

DETAILED DESCRIPTION:
This is a multi-national, multi-center, fixed-dose, 52-week, open-label extension study. After completing participation in either RETHINK-ALZ (PTI-125-06) or REFOCUS-ALZ (PTI-125-07), subjects will have the option to participate in this study. After the subject provides consent and the Investigator confirms the subject satisfies both inclusion and exclusion criteria, the study drug will be administered at the research site on Study Day 1 and subsequent visits will be scheduled.

We anticipate up to 1600 subjects may enroll in this study. Approximately up to 150 clinical sites in the USA, Canada, South Korea, and Australia will have the option to participate in this collaborative research effort.

For subjects electing to participate, the clinical and laboratory assessments from the Week 76 (REFOCUS-ALZ) or Week 52 (RETHINK-ALZ) End-of-Treatment visit will serve as Baseline Visit assessments for the open-label study on Study Day 1. All subjects will return in 4 weeks and every 12 weeks thereafter for safety assessments. At all post-baseline visits, subjects will report any adverse events since their last visit. In addition to adverse event monitoring, safety will be evaluated at every visit by vital signs, brief examinations, clinical laboratory tests (biochemistry, hematology, and urinalysis) and the Columbia Suicide Severity Rating Scale (C-SSRS). Study drug use since the last visit will be assessed and a new bottle of study drug will be dispensed.

The emerging subject safety assessments will be monitored throughout the study by an independent Data Safety Monitoring Board (DSMB).

ELIGIBILITY:
Inclusion Criterion:

* Completed RETHINK-ALZ (PTI-125-07) or REFOCUS-ALZ (PTI-125-06).
* Clinical presentation continues to be consistent with Alzheimer's disease.
* Availability of a study partner.

Exclusion Criteria:

* Residence in a skilled nursing facility requiring 24-hour care.
* Evidence of a neurologic condition other than AD that significantly contributes to the subject's dementia.
* Current clinically significant psychiatric diagnosis other than AD.
* Unstable, clinically significant medical condition other than AD.
* Any medical condition that in the opinion of the investigator may affect safety or ability to complete the study.

Ages: 51 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1081 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Kupiec, MD, Study Director — Cassava Sciences, Inc.
Locations (133):
- United States (106):
  - MDFirst Research, Chandler, Arizona
  - CCT Research - Gilbert Neurology Partners, Gilbert, Arizona
  - Xenoscience, Inc., Phoenix, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - North County Neurology Associates, Carlsbad, California
  - Axiom Research, LLC, Colton, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Neuro-Pain Medical Center, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Sun Valley Research Center, Inc., Imperial, California
  - Senior Clinical Trials, Laguna Hills, California
  - Shankle Clinic and Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Pacific Research Network, LLC, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Mountain Neurological Research Center, Basalt, Colorado
  - Colorado Neurological Research Center, PC, Denver, Colorado
  - Ki Health Partners, LLC, Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Neurology Offices of South Florida, Boca Raton, Florida
  - K2 Medical Research- Ocoee, Clermont, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Galiz Research, Hialeah, Florida
  - Infinity Clinical Research - Sunrise, Hollywood, Florida
  - Luminous Clinical Research, Homestead, Florida
  - CNS Healthcare - Jacksonville, Jacksonville, Florida
  - Charter Research, Lady Lake, Florida
  - ClinCloud, Maitland, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Central Miami Medical Institute (GMI), Miami, Florida
  - Mind Institute at Miami Jewish Health, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Brainstorm Research, Miami, Florida
  - South Florida Research Phase I-IV INC, Miami Springs, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Health Synergy Clinical Research, Okeechobee, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - Medical Research, Port Orange, Florida
  - Intercoastal Medical Group - Sarasota, Sarasota, Florida
  - Alzheimer's Research & Treatment Center, Stuart, Florida
  - Clinical Research of Brandon, LLC (Tampa), Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Alzheimer's Research & Treatment Center, Wellington, Florida
  - Premier Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Charter Research, Winter Park, Florida
  - Columbus Memory Center, PC, Columbus, Georgia
  - Accel Research Sites - NeuroStudies, Decatur, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Advocate Aurora Health - Advocate Memory Center, Park Ridge, Illinois
  - Ascension Via Christi Research, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Neuro Medical Clinic of Central Louisiana, LLC, Alexandria, Louisiana
  - Neurology Center of New England, Foxborough, Massachusetts
  - ActivMed Practices & Research, LLC, Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Boston Neuro Research Center, North Dartmouth, Massachusetts
  - Headlands Eastern MA LLC, Plymouth, Massachusetts
  - MedVadis Research, Waltham, Massachusetts
  - Clinical Research Professionals, Chesterfield, Missouri
  - CCT Research - Papillion Research Center, Papillion, Nebraska
  - Patient First MD, Middletown, New Jersey
  - Advanced Clinical Institute, Inc, Neptune City, New Jersey
  - Global Medical Institutes, LLC, Princeton, New Jersey
  - The Cognitive and Research Center of New Jersey (CRCNJ), Springfield, New Jersey
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Neurology Specialists of Monmouth County, West Long Branch, New Jersey
  - Albuquerque Neuroscience, Inc, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Neurological Associates of Albany, Albany, New York
  - Dent Neurologic Institute, Amherst, New York
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - SPRI Clinical Trials Brooklyn, Brooklyn, New York
  - Velocity Clinical Research, Formerly Clarity Clinical Research, East Syracuse, New York
  - Parker Jewish Institute for Health Care & Rehabilitation, New Hyde Park, New York
  - Mid Hudson Medical Research, New Windsor, New York
  - NY Neurology Associates, New York, New York
  - University of Rochester Medical Center - Alzheimer's Disease Care, Research and Education Program, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Triad Clinical Trials, LLC, Greensboro, North Carolina
  - Alzheimer's Memory Center, Matthew, North Carolina
  - Accellacare Research of Winston-Salem, Winston-Salem, North Carolina
  - Insight Clinical Trials LLC, Beachwood, Ohio
  - NeuroScience Research Center, LLC, Canton, Ohio
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - the Ohio State University, Columbus, Ohio
  - Neurology Diagnostics, Dayton, Ohio
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Summit Research Network, LLC, Portland, Oregon
  - Center for Cognitive Health - Portland, Portland, Oregon
  - Keystone Clinical Studies, LLC, Plymouth Meeting, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Palmetto Clinical Research, Summerville, South Carolina
  - Senior Adults Specialty Research, Inc, Austin, Texas
  - Texas Neurology, PA, Dallas, Texas
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Mt. Olympus Medical Research, LLC, Katy, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Re:Cognition Health, Fairfax, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Memory and Brain Wellness Center at Harborview, Seattle, Washington
- Australia (7):
  - KaRa Institute of Neurological Diseases Pty. Ltd., Macquarie Park, New South Wales
  - The University of Queensland, Herston, Queensland
  - Delmont Consulting Suites, Glen Iris, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Eastern Health, Melbourne, Victoria
  - Alzheimer's Research Australia, Nedlands, Western Australia
- Canada (12):
  - OCT Research ULC DBA Okanagan Clinical Trials, Kelowna, British Columbia
  - Dr. George Dumont University Hospital Centre, Moncton, New Brunswick
  - True North Clinical Research - Halifax/Nova Scotia, Halifax, Nova Scotia
  - True North Clinical Research - New Minas, New Minas, Nova Scotia
  - St. Joseph's Health Care London, London, Ontario
  - Ottawa Memory Clinic, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - The Centre for Memory and Aging, Toronto, Ontario
  - Q & T Research, Sherbrooke, Quebec
  - Diex Research - Sherbrooke, Sherbrooke, Quebec
  - Alpha Recherche Clinique, Québec
- Puerto Rico (3):
  - Barbara Diaz Hernandez Md Research, Inc., San Juan, PR
  - Santa Cruz Behavioral PSC, Bayamón
  - Inspira Clinical Research, San Juan
- South Korea (5):
  - Kyungpook National University Chilgok Hospital, Daegu, Buk-gu
  - Chonnam National University Hospital, Gwangju, Dong-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Hospital, Namyangju, Incheon
  - Inha Unviersity Medical Center, Incheon, Jung-gu

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label extension study.
Period: Overall Study
Arm/Group | Simufilam 100 mg
Started (First participant in study November 07, 2022) | 1081
Completed | 300
Not Completed | 781
Not completed — Adverse Event | 24
Not completed — Death | 7
Not completed — Lost to Follow-up | 16
Not completed — Non-Compliance | 3
Not completed — Physician Decision | 6
Not completed — Sponsor Requests to be Withdrawn | 7
Not completed — Withdrawal by Subject | 71
Not completed — Study Terminated by Sponsor | 630
Not completed — Other | 17

BASELINE CHARACTERISTICS:
Population: 1079 participants are in the safety analysis (with baseline characteristics).
Arm/Group | Simufilam
Number analyzed (Participants) | 1079
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 144
  >=65 years | 935
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 583
  Male | 496
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 87
  Not Hispanic or Latino | 977
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 45
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 54
  White | 962
  More than one race | 1
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  Canada | 115
  Puerto Rico | 7
  South Korea | 22
  United States | 890
  Australia | 45
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.59 (6.892)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: To evaluate the long-term safety and tolerability of simufilam 100 mg tablets in subjects who have completed one of the two double-blind simufilam phase 3 studies.
Time Frame: Baseline to 52 weeks
Population: The number of subjects in the analysis (1079) differs by two subjects compared to the Participant Flow module (1081), because there are two subjects who were enrolled but did not receive study treatment and were not included in the Safety Analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- Simufilam 100mg: simufilam 100 mg oral tablet, twice daily
Arm/Group | Simufilam 100mg
Number analyzed (Participants) | 1079
Participants
  Number of subjects with mild AEs | 299
  Number of subjects with moderate AEs | 198
  Number of subjects with severe AEs | 63
  Number of subjects with no AEs | 519

ADVERSE EVENTS:
Time Frame: Up to 54 weeks after subjects took their first dose of study drug, or until resolution or stabilization of any AEs ongoing at the end of the study.
Arm/Group | Simufilam 100mg
All-Cause Mortality (participants affected / at risk) | 9/1079
Serious Adverse Events (participants affected / at risk) | 92/1079
Other Adverse Events (participants affected / at risk) | 0/1079
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simufilam 100mg (N=1079)
Syncope (Nervous system disorders) | 10 (10)
Cerebrovascular accident (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 2 (2)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Dementia Alzheimer's Type (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7)
Urinary tract infection (Infections and infestations) | 4 (4)
COVID-19 (Infections and infestations) | 3 (3)
Diverticulitis (Infections and infestations) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Myocardial infarction (Cardiac disorders) | 3 (3)
Coronary artery disease (Infections and infestations) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (2)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural constipation (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemotoma (Injury, poisoning and procedural complications) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Gastrointestinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2)
Mental status changes (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Hallucinations, mixed (Psychiatric disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Gait inability (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostrate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and PI must request review and comment of any proposed publication by the sponsor at least 90 days prior to submission of the publication. The sponsor will advise of any information which is confidential information or which may impair the sponsor's ability to obtain patent protection, and has the right to require confidential information or factual errors to be removed, or to delay the proposed publication by an additional 90 days to allow the sponsor to seek patent protection.

DOCUMENTS (2):
  • Study Protocol (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT05575076/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT05575076/SAP_001.pdf